CLINICAL TRIAL: NCT01122758
Title: (COPD History Assessment In SpaiN): "Estudio Sobre la Evolución Multidimensional de la Enfermedad Pulmonar Obstructiva Crónica (EPOC)".
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) History Assessment In SpaiN (CHAIN)
Acronym: CHAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cimera (Network)
Responsible Party: Dr Ciro Casanova, Hospital Universitario Nuestra Señora de la Candelaria
Other Study IDs: CHAIN; IB1323/10PI (Other: CEIC Illes Balears)
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: COPD
Keywords: Cohort; COPD; Natural history; Phenotyping; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — complete blood and serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD cohort: Inclusion criteria:
  * Patients ≥ 35 years.
  * Diagnosis of COPD (GOLD PBD FEV1/FVC ratio <0.70).
  * Being in a stable phase of disease (8 weeks without exacerbation).
  * Cummulative smoking ≥ 10 pack-years.
  * Absence of asthma or other chronic respiratory disease that justify the ventilatory disorder (although a history of asthma is not an exclusion criteria);
  * Absence of malignancy or very serious comorbidities that would prevent study completion.
  Exclusion criteria:
  * Patients <35 years.
  * Recent exacerbation (<8 weeks).
  * Not giving written informed consent.
  * Presence of asthma or other chronic respiratory disease justifying the ventilatory disorder,
  * Diffuse bronchiectasis not associated with COPD.
  * Presence of malignancy or very serious comorbidities that would prevent study completion.
  * Difficulty to perform appropriate follow-up.
- Control cohort: Inclusion criteria:
  * Patients ≥ 35 years.
  * Absence of diagnosis of COPD (GOLD PBD FEV1/FVC ratio >=0.70).
  * Cummulative smoking ≥ 10 pack-years.
  * Absence of asthma or other chronic respiratory disease that justify the ventilatory disorder (although a history of asthma is not an exclusion criteria);
  * Absence of malignancy or very serious comorbidities that would prevent study completion.
  Exclusion criteria:
  * Patients <35 years.
  * Not giving written informed consent.
  * Presence of asthma or other chronic respiratory disease justifying the ventilatory disorder,
  * Diffuse bronchiectasis not associated with COPD.
  * Presence of malignancy or very serious comorbidities that would prevent study completion.
  * Difficulty to perform appropriate follow-up.

SUMMARY:
The research project CHAIN (COPD Assessment History in Spain): "A Multidimensional Study on the Evolution of Chronic Obstructive Pulmonary Disease (COPD)is a multicentre, observational study conducted in several areas of Spain aimed to better define COPD natural history and its phenotypes

DETAILED DESCRIPTION:
Observational studies are needed to ascertain the natural history and progression of COPD, and to better define its phenotypes. These two aspects are considered fundamental to a proper evaluation of current (and future) COPD treatment options, and it could possibly justify the limited impact of recent major drug trials.

Currently, there remain gaps in the natural history of patients with COPD. Most data are from analysis of mild COPD patients or smokers, usually measuring only fall in FEV1, and both have significant limitations in design and interpretation.

Studies in more severe patients with COPD have also been conducted mainly by studying lung function, possibly influenced by the recommendations of current guidelines for disease management. In recent years, we have more longitudinal data on changes in exercise capacity, imaging, and biomarkers, among other variables of interest, but our knowledge is yet partial.

The research project CHAIN (COPD Assessment History in Spain): "A Multidimensional Study on the Evolution of Chronic Obstructive Pulmonary Disease (COPD) is a multicenter observational study that will follow prospectively two cohorts: a) a COPD group active or former smokers (COPD cohort) and b) a group of active smokers or former smokers without COPD (control cohort). Both cohorts will be followed up for a period of at least 5 years, with visits every 12 months (and phone controls at least every 6 months). We will try to extend the monitoring of the cohort up to 10 years. CHAIN is supported by the PII of COPD SEPAR

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 35 years.
* Diagnosis of COPD (GOLD PBD FEV1/FVC ratio <0.70).
* Being in a stable phase of disease (8 weeks without exacerbation).
* Cummulative smoking ≥ 10 pack-years.
* Absence of asthma or other chronic respiratory disease that justify the ventilatory disorder (although a history of asthma is not an exclusion criteria);
* Absence of malignancy or very serious comorbidities that would prevent study completion.

Exclusion Criteria:

* Patients <35 years.
* Recent exacerbation (<8 weeks).
* Not giving written informed consent.
* Presence of asthma or other chronic respiratory disease justifying the ventilatory disorder,
* Diffuse bronchiectasis not associated with COPD.
* Presence of malignancy or very serious comorbidities that would prevent study completion.
* Difficulty to perform appropriate follow-up.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the outpatient clinics, pulmonary function labs, and / or pulmonology wards of each participating center
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2009-12; Primary Completion 2014-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
To better determine COPD with a multidimensional assessment and the phenotypic progression of COPD | 5 years

SECONDARY OUTCOMES:
- Progression of the disease by degree of severity. - Effect of treatment on disease progression and variability of response according to phenotypes. - Geographical differences. - The impact of exacerbations. - The importance of comorbidities and | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Casanova, MD, Principal Investigator — Hospital Nuestra Señora de la Candelaria
Locations (2):
- Spain (2):
  - Ciro Casanova, Santa Cruz de Tenerife, Canary Islands
  - 40-50 additional centres throughout Spain, Bunyola

REFERENCES:
- [Derived] Casanova C, Gonzalez-Davila E, de Torres JP, Cabrera C, Cosio BG, O'Donnel DE, Martinez-Gonzalez C, Solanes I, Fuster A, Gotera C, Marin A, Amado C, Iscar M, Marin JM, Neder JA, Feu N, Soriano JB, Lopez-Campos JL, Divo M, Peces-Barba G, Celli BR. Lung Diffusing Capacity Improves the Prognostic Validity of the GOLD Spirometric Staging in COPD. Arch Bronconeumol. 2026 Jan;62(1):20-27. doi: 10.1016/j.arbres.2025.05.004. Epub 2025 May 16. English, Spanish. PMID 40447521
- [Derived] Casanova C, Gonzalez-Davila E, Martinez-Gonzalez C, Cosio BG, Fuster A, Feu N, Solanes I, Cabrera C, Marin JM, Balcells E, Peces-Barba G, de Torres JP, Marin-Oto M, Calle M, Golpe R, Ojeda E, Divo M, Pinto-Plata V, Amado C, Lopez-Campos JL, Celli BR. Natural Course of the Diffusing Capacity of the Lungs for Carbon Monoxide in COPD: Importance of Sex. Chest. 2021 Aug;160(2):481-490. doi: 10.1016/j.chest.2021.03.069. Epub 2021 Apr 18. PMID 33878339
- [Derived] Calle Rubio M, Rodriguez Hermosa JL, de Torres JP, Marin JM, Martinez-Gonzalez C, Fuster A, Cosio BG, Peces-Barba G, Solanes I, Feu-Collado N, Lopez-Campos JL, Casanova C; CHAIN Study Investigators. COPD Clinical Control: predictors and long-term follow-up of the CHAIN cohort. Respir Res. 2021 Feb 4;22(1):36. doi: 10.1186/s12931-021-01633-y. PMID 33541356
- [Derived] Soriano JB, Hahsler M, Soriano C, Martinez C, de-Torres JP, Marin JM, de Lucas P, Cosio BG, Fuster A, Casanova C; CHAIN investigators. Temporal transitions in COPD severity stages within the GOLD 2017 classification system. Respir Med. 2018 Sep;142:81-85. doi: 10.1016/j.rmed.2018.07.019. Epub 2018 Aug 3. PMID 30170807
- [Derived] Martinez-Gonzalez C, Casanova C, de-Torres JP, Marin JM, de Lucas P, Fuster A, Cosio BG, Calle M, Peces-Barba G, Solanes I, Aguero R, Feu-Collado N, Alfageme I, Romero Plaza A, Balcells E, de Diego A, Marin Royo M, Moreno A, Llunell Casanovas A, Galdiz JB, Golpe R, Lacarcel Bautista C, Cabrera C, Marin A, Soriano JB, Lopez-Campos JL; CHAIN Study Investigators. Changes and Clinical Consequences of Smoking Cessation in Patients With COPD: A Prospective Analysis From the CHAIN Cohort. Chest. 2018 Aug;154(2):274-285. doi: 10.1016/j.chest.2018.02.007. Epub 2018 Feb 22. PMID 29476876
- [Derived] Cosio BG, Soriano JB, Lopez-Campos JL, Calle-Rubio M, Soler-Cataluna JJ, de-Torres JP, Marin JM, Martinez-Gonzalez C, de Lucas P, Mir I, Peces-Barba G, Feu-Collado N, Solanes I, Alfageme I, Casanova C; CHAIN Study. Defining the Asthma-COPD Overlap Syndrome in a COPD Cohort. Chest. 2016 Jan;149(1):45-52. doi: 10.1378/chest.15-1055. Epub 2016 Jan 6. PMID 26291753
- [Derived] Casanova C, Marin JM, Martinez-Gonzalez C, de Lucas-Ramos P, Mir-Viladrich I, Cosio B, Peces-Barba G, Solanes-Garcia I, Aguero R, Feu-Collado N, Calle-Rubio M, Alfageme I, de Diego-Damia A, Irigaray R, Marin M, Balcells E, Llunell A, Galdiz JB, Golpe R, Lacarcel C, Cabrera C, Marin A, Soriano JB, Lopez-Campos JL, Soler-Cataluna JJ, de-Torres JP; COPD History Assessment in Spain (CHAIN) Cohort. Differential Effect of Modified Medical Research Council Dyspnea, COPD Assessment Test, and Clinical COPD Questionnaire for Symptoms Evaluation Within the New GOLD Staging and Mortality in COPD. Chest. 2015 Jul;148(1):159-168. doi: 10.1378/chest.14-2449. PMID 25612228
- [Derived] de Torres JP, Marin JM, Martinez-Gonzalez C, de Lucas-Ramos P, Mir-Viladrich I, Cosio B, Peces-Barba G, Calle-Rubio M, Solanes-Garcia I, Aguero Balbin R, de Diego-Damia A, Feu-Collado N, Alfageme Michavila I, Irigaray R, Balcells E, Llunell Casanovas A, Galdiz Iturri JB, Marin Royo M, Soler-Cataluna JJ, Lopez-Campos JL, Soriano JB, Casanova C; COPD History Assessment in Spain (CHAIN) Cohort*. Clinical application of the COPD assessment test: longitudinal data from the COPD History Assessment in Spain (CHAIN) cohort. Chest. 2014 Jul;146(1):111-122. doi: 10.1378/chest.13-2246. PMID 24522636
- See also: SEPAR-Sociedad Española de Neumología y Cirugía Torácica — http://www.separ.es